CLINICAL TRIAL: NCT06863064
Title: Exploring the Effects of Perioperative Dexmedetomidine on the Incidence of Postoperative Delirium, Acute and Chronic Pain, and Sleep Quality in Patients Undergoing Brain Tumor Surgery
Brief Title: Brain Tumor Surgery and Postoperative Delirium
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KMUHIRB-F(I)-20240297
Record Dates: First submitted 2025-02-04; First posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Brain Tumor
Keywords: brain tumor; postoperative delirium
MeSH Terms: conditions — Brain Neoplasms; Emergence Delirium | interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participant Group (Experimental): brain tumor postoperative
  Interventions: Drug: Dexmedetomidine; Drug: Normal Saline

INTERVENTIONS:
Drug: Dexmedetomidine — During the surgery, target-controlled infusion (TCI) pumps were used, employing the Dyck model for continuous infusion of propofol, with the target plasma concentration maintained at 0.2 ng/ml. Postoperatively, propofol was infused at a rate of 0.2-0.4 mcg/kg/hr according to the intensive care unit's protocol, until the patient had the endotracheal tube removed.
Drug: Normal Saline — During the surgery, equal volumes of saline were injected. After the surgery, the patient was transferred to the intensive care unit, where propofol was continuously infused at a rate of 0.2-0.4 mcg/kg/hr according to the ICU protocol, until the endotracheal tube was removed.

SUMMARY:
1. To explore whether the combined administration of dexmedetomidine during and after surgery in patients undergoing brain tumor resection is an effective and safe modality to prevent postoperative delirium and improve sleep quality than giving it alone after surgery.
2. To explore whether intraoperative and postoperative administration of dexmedetomidine to patients undergoing brain tumor surgery can reduce postoperative acute pain and prevent chronic pain.
3. To explore whether intraoperative and postoperative administration of dexmedetomidine to patients undergoing brain tumor surgery can provide stable anesthesia depth, hemodynamics and reduce the dose of anesthetics, thereby accelerating patient recovery.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old and less than 80 years old
* receive brain tumor surgery with ASA II~III.

Exclusion Criteria:

* under the age of 18 or over 80
* consciousness unclear
* those who have not signed a consent form
* those with high anesthesia risk ASA IV or higher

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment and Documentation of Delirium | Perioperative
  Confusion assessment method in intensive care unit using questionnaire(CAM-ICU), The evaluation method is "yes" or "no," with "no" being the best.
Assessment and Documentation of Delirium | Perioperative
  3-minute diagnostic interview with confusion assessment method (3D-CAM), The evaluation method is "yes" or "no," with "no" being the best.
Assessment and Documentation of Delirium | Perioperative
  Richmond Agitation-Sedation Scale (RASS) ,The score ranges from +4 to -5, with +4 being the best.
Assessment and Documentation of Delirium | 1 to 3 days post-surgery.
  Numerical Rating Scale (NRS) ,The score ranges from 0 to 10, with 0 being the best.
Assessment and Documentation of Delirium | 1 to 3 days post-surgery.
  Richards Campbell Sleep Questionnaire (RCSQ) ,The score ranges from 0 to 100, with 100 being the best.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Taiwan